CLINICAL TRIAL: NCT02551575
Title: Efficacy and Safety of Qingre Huoxue Comprehensive Therapy in the Treatment of Rheumatoid Arthritis (RA): A Randomized, Double-blind, Double-dummy, Multi-center Trial
Brief Title: Efficacy and Safety of Traditional Chinese Medicine (TCM) Comprehensive Therapy in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Quan Jiang, Director，Devision of Rheumatology, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013BAI02B06
Record Dates: First submitted 2015-08-26; First posted 2015-09-16 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment of MTX and HCQ (Active Comparator): Patients were treated with methotrexate (MTX), hydroxychloroquine (HCQ), oral Qingre Huoxue granule placebo and Qingre Huoxue external preparation placebo.
  Interventions: Drug: Treatment of MTX and HCQ
- Treatment of TCM (Experimental): Patients were treated with oral Qingre Huoxue granule, Qingre Huoxue external preparation, methotrexate placebo and hydroxychloroquine placebo.
  Interventions: Drug: Treatment of TCM
- Integrative Medicine (Experimental): The patients were treated with methotrexate, hydroxychloroquine, oral Qingre Huoxue granule and Qingre Huoxue external preparation.
  Interventions: Drug: Integrative Medicine

INTERVENTIONS:
Drug: Treatment of MTX and HCQ — Methotrexate: 10-15mg per week according to patient's weight, oral, for 24 weeks.
  Hydroxychloroquine: 200mg, 2 times a day, oral, for 24 weeks. Qingre Huoxue granule placebo: 10g, 2 times a day, oral, for 24 weeks. Qingre Huoxue external preparation placebo: 20g, 1 times a day, external, for 4 weeks, then 10g, 1 times a day, external, for 8 weeks.
  Other Names: Treatment of MTX, HCQ and Qingre Huoxue placebo
  Arms: Treatment of MTX and HCQ
Drug: Treatment of TCM — Qingre Huoxue granule: 10g, 2 times a day, oral, for 24 weeks. Qingre Huoxue external preparation: 20g, 1 times a day, external, for 4 weeks, then 10g, 1 times a day, external, for 8 weeks.
  Methotrexate placebo: 10-15mg per week according to patient's weight, oral, for 24 weeks.
  Hydroxychloroquine placebo: 200mg, 3 times a day, oral, for 24 weeks.
  Other Names: Qingre Huoxue medicines，MTX placebo and HCQ placebo
  Arms: Treatment of TCM
Drug: Integrative Medicine — Qingre Huoxue granule: 10g, 2 times a day, oral, for 24 weeks. Qingre Huoxue external preparation: 20g, 1 times a day, external, for 4 weeks, then 10g, 1 times a day, external, for 8 weeks.
  Methotrexate: 10-15mg per week according to patient's weight, oral, for 24 weeks.
  Hydroxychloroquine: 200mg, 3 times a day, oral, for 24 weeks.
  Other Names: Treatment of Qingre Huoxue medicines，MTX and HCQ
  Arms: Integrative Medicine

SUMMARY:
This is prospective randomized, controlled study to evaluate the efficacy and safety of Qingre Huoxue comprehensive therapy in treating of patients with early Rheumatoid Arthritis (RA). The major outcome index is the change from baseline to week 24 in Disease Activity Score (DAS28), and minor outcome indexes include American College of Rheumatology (ACR)20/50/70, PRO score, Sharp score and OMERACT RAMRIS score. The adverse events at any time were recorded to evaluate the safety.

DETAILED DESCRIPTION:
Three arms were included in this study, and treatment with MTX and HCQ is defined as active comparator. Treatment of TCM，including Qingre Huoxue granule, Qingre Huoxue external preparation, MTX placebo and HCQ placebo, is defined as one experimental arm. Treatment of integrative medicine，including Qingre Huoxue granule, Qingre Huoxue external preparation, MTX and HCQ, is defined as another experimental arm.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rheumatoid arthritis as determined by the 1987 ACR classification criteria.
* Diagnosed with TCM dampness heat and blood stasis syndrome
* The course of RA is not more than 5 years.
* Swollen joint (SJC)≥2 and tender joint count(TJC)≥3.
* Erythrocyte Sedimentation Rate（ESR）≥20 mm/hr
* Patients who take disease-modifying antirheumatic drugs for at least 3 months on a stable dose, and retain the same treatment during the study.
* Age 18-65 years with informed consent

Exclusion Criteria:

* Patients with skin burst or allergies.
* Patients with cancer or other malignant disease such as cardiovascular, hematopoietic, liver and kidney disease, and psychopath
* Active or chronic infection, including HIV, hepatitis C virus, hepatitis B virus, tuberculosis
* Previous treated with tripterygii, glucocorticoid or biologic disease-modifying antirheumatic drug (DMARD) in 3 months.
* Previous treated with MTX or HCQ
* Patients with retinopathy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The change from Baseline to week 24 in Disease Activity Score (DAS28) | 0 weeks, 12 weeks, 24 weeks
  Disease Activity Score for 28-joint counts was based on the erythrocyte sedimentation rate(ESR) (DAS28-4[ESR])

SECONDARY OUTCOMES:
The proportion of patients achieving ACR20/50/70 | 0 week, 12 weeks, 24 weeks
  ACR20/50/70 is referred to American College of Rheumatology Criteria.
The change from baseline to week 24 in the score on the patient report outcome (PRO) | 0 week, 12 weeks, 24 weeks
  PRO scores ranges from 0 to 3, with higher scores indicating greater disability
The change in Sharp score | 0 week, 52 weeks
  The change in X-Ray from baseline to week 52.
The change in OMERACT RAMRIS score | 0 week, 24 weeks
  The change in Magnetic Resonance Imaging from baseline to week 24.
The number of adverse events | 24 weeks
  The number of adverse events that are related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Quan, MD, Study Director — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Gong X, Liu WX, Tang XP, Wang J, Liu J, Huang QC, Liu W, Fang YF, He DY, Liu Y, Gao ML, Wu QJ, Chen S, Li ZB, Wang Y, Xie YM, Zhang JL, Zhou CY, Ma L, Wang XC, Zhang C, Jiang Q. Traditional Chinese Medicine Qingre Huoxue Treatment vs. the Combination of Methotrexate and Hydroxychloroquine for Active Rheumatoid Arthritis: A Multicenter, Double-Blind, Randomized Controlled Trial. Front Pharmacol. 2021 May 25;12:679588. doi: 10.3389/fphar.2021.679588. eCollection 2021. PMID 34113254